CLINICAL TRIAL: NCT01495312
Title: 24-hr Intraocular Pressure (IOP) Patterns of Glaucoma Patients After Selective Laser Trabeculoplasty (SLT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to staff departures unable to execute this study so requested closure. There were no study procedures performed & no participants enrolled.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Eunice Williams-Steppe, Research Associate, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TFSLT1
Record Dates: First submitted 2011-12-12; First posted 2011-12-20 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Glaucoma
Keywords: IOP fluctuations; during two 24-hour periods
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SLT (Experimental)
  Interventions: Device: SLT (selective laser trabeculoplasty ) SENSIMED Triggerfish

INTERVENTIONS:
Device: SLT (selective laser trabeculoplasty ) SENSIMED Triggerfish — SLT (single session; 180 to 360 degrees of angle will be treated)

SUMMARY:
The purpose of this study is to determine the relationship between Intraocular Pressure (IOP) fluctuations of glaucoma patients as recorded with an IOP-sensing contact lens (SENSIMED Triggerfish®), during two 24-hour periods after selective laser trabeculoplasty (SLT) for routine treatment of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must correspond to all other inclusion criteria in order to be eligible for the investigation.

  * Subject is able to comply with the study procedures
  * 18-80 years old
  * Subjects diagnosed with glaucoma, based on presence of repeatable visual field loss and/or glaucomatous optic neuropathy based on masked review of optic disc stereophotographs and under ocular hypotensive treatment, or diagnosed with ocular hypertension, with an IOP of > 22 mmHg at the screening visit and under ocular hypotensive treatment.
  * Subject has consented to be in the trial
  * Visual acuity of 20/200 or better
  * Ability to understand the character and individual consequences of the study
  * For women of childbearing potential, adequate contraception

Exclusion Criteria:

* Subjects presenting with any of the following criteria will not be included in the trial:

  * Subjects with contraindications for wearing contact lenses
  * Severe dry eye syndrome
  * Keratoconus or other corneal abnormality
  * Conjunctival or intraocular inflammation
  * Eye surgery prior to and throughout the study.
  * Full frame metal glasses during SENSIMED Triggerfish® monitoring
  * Known hypersensitivity to silicone, plaster or ocular anesthesia (proparacaine)
  * Pregnancy and lactation
  * Simultaneous participation in other clinical studies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Estimated); Study Completion 2013-08-12 (Actual)

PRIMARY OUTCOMES:
IOP | 2 months after SLT

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, La Jolla, California, United States